CLINICAL TRIAL: NCT07213908
Title: Comparing Two School-Based Sleep Health Interventions To Promote Sleep Quality in Youth
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Collaborators: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Lauren Asarnow, Medical Staff/USC Faculty CWR • Neurology CWR, Children's Hospital Los Angeles
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: APP-25-03648; SL-2024C1-37532-IC (Other: PCORI)
Record Dates: First submitted 2025-09-29; First posted 2025-10-09 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Sleep
Keywords: Adolescents; Sleep; Schools; Cognitive Behavioral Sleep Intervention

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sleep Health Education (SHE) (Active Comparator): Participants will be given access to a program, developed for the proposed project, with American Academy of Sleep Medicine (AASM) videos, worksheets and sleep diaries aimed to improve sleep health.
  Interventions: Behavioral: Sleep Health Education (SHE)
- Transdiagnostic Sleep and Circadian intervention (TS-C-STEP (Experimental): In the TS-C-STEP condition, all participants initially are given access to the TS-C program. TS-C is an evidence based cognitive behavioral sleep intervention. Youth will be stepped up to higher levels of care dependent on their progress with the program.
  Interventions: Behavioral: TS-C-STEP

INTERVENTIONS:
Behavioral: TS-C-STEP — Cognitive behavioral sleep intervention.
  Arms: Transdiagnostic Sleep and Circadian intervention (TS-C-STEP
Behavioral: Sleep Health Education (SHE) — Health Education
  Arms: Sleep Health Education (SHE)

SUMMARY:
The goal of this clinical trial is to conduct a comparative effectiveness trial that will evaluate two school-based interventions to improve adolescent sleep health: the standard Sleep Health Education (SHE) and a stepped care version of the Transdiagnostic Sleep and Circadian intervention (TS-C-STEP). The main questions it aims to answer [is/are]:

* TS-C-STEP will yield superior outcomes relative to SHE at post-treatment and up to 12 months following treatment.
* In this large and diverse sample, vulnerable subgroups (e.g. socioeconomically disadvantaged, racial, ethnic, rural, and youth with comorbid learning and/or mental health conditions) will experience greater benefits from TS-C-STEP compared to SHE on primary and secondary outcomes.

Researchers will compare sleep quality to determine which intervention is most effective.

ELIGIBILITY:
Inclusion Criteria:

* Age 12-18 years old
* Sleep health problem (i.e. insomnia, evening circadian preference, short sleep duration, poor sleep quality)
* Able to participate in a general education classroom.

Exclusion Criteria:

* Previous participation in the study;
* Symptoms or illness that precludes informed consent or engagement in study procedures ; youth not fluent in English, parent not fluent in English, or Spanish.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1320 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2030-02-01 (Estimated); Study Completion 2030-06-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline for total score sleep quality using the Pittsburgh Sleep Quality Index. | Baseline to 14 months
  A self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval. The sum of scores yields one global score with a minimum score of 0 and a maximum score of 21. A higher score indicates more self-reported sleep problems.

SECONDARY OUTCOMES:
Change from baseline for total insomnia severity score sleep health using the insomnia severity index. | Baseline to 14 months
  7-item scale assessing the perceived severity of insomnia symptoms. The sum of scores yields a total score with a minimum score of 0 and a maximum score of 28. A higher score indicates more severe insomnia symptoms.
Change from baseline for total evening circadian preference score sleep health using the Children's Morningness and Eveningness Preference. | Baseline to 14 months
  Evening Circadian Preference is a reliable and valid 10-item measure of circadian preference among youth
Change from baseline for total sleep related impairment score sleep health using the PROMIS sleep related impairment questionnaire. | Baseline to 14 months
  PROMIS is a well-validated 8-item measure which assesses self-reported perceptions of alertness, sleepiness, and tiredness during usual waking hours, and the perceived functional impairments during wakefulness associated with sleep problems or impaired alertness. A total raw score can range from 8 to 40, with a higher score indicating more sleep related impairment.
Change from baseline for sleep duration estimates from sleep diaries. | Baseline to 14 months
  Sleep diary asks participants about daily morning estimates of sleep the night prior parameters yield a reliable and valid clinical index of self-reported sleep duration.
Change from baseline for quality of life and functioning using the PROMIS Global Health Questionnaire. | Baseline to 14 months
  The PROMIS Scale Global Health is a ten-item patient reported measure of physical, mental and social health.
Change from baseline for academic functioning using official transcripts provided by participants. | Baseline to 14 months
  Academic Functioning Youth participants will be asked to provider their official academic transcripts.
Change from baseline for overall mental health using your self-report (youth) | Baseline to 14 months
  Youth Self-Report (YSR) is a widely used self-report measure that assesses problem behaviors across multiple domains and provides a summary of total problems which can range from 0 to 224 in raw scores; a higher score indicates more self-reported problems. Raw scores are converted to standardized T-scores, which are adjusted for age and gender and are used to compare a youth's score to a normative sample.
Change from baseline for overall mental health using child-behavior checklist (parent). | Baseline to 14 months
  Child Behavior Checklist (CBCL) completed by parents is a widely used child-report measure that assesses problem behaviors across multiple domains and provides a summary of total problems which can range from 0 to 198 in raw scores; a higher score indicates more self-reported problems. Raw scores are converted to standardized T-scores, which are adjusted for age and gender and are used to compare a youth's score to a normative sample.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Asarnow,, PhD, Principal Investigator — Children's Hospital Los Angeles
Locations (2):
- United States (2):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Nationwide Children's Hospital, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol